CLINICAL TRIAL: NCT01912846
Title: An Interactive Advance Care Planning Intervention to Facilitate a Good Death for Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Siew Tzuh Tang, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HMRPD1C0011; NHRI-EX102-10208PI (Other Grant/Funding Number: National Health Research Institute, Taiwan)
Record Dates: First submitted 2013-07-18; First posted 2013-07-31 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: End Stage Cancer
Keywords: End-of-life care; Preference of end-of-life care; RCT; Terminally ill cancer patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention usual care intervention (Sham Comparator): Interventions includes prognosis disclosure and discussions of EOL care as needed as in current clinical practices.
  Interventions of the attention usual care arm include a consistent master prepared nurse on the study team will provide the attention portion of the care and a workbook and a video with educational materials. The initial meeting will occur before the patient discharges from hospital and the usual care nurse will give patients and family caregivers a workbook and a video with educational materials on how to manage common symptoms and a comprehensive list of resources available, including patient support organizations, support and financial assistance through the social work department.
  Interventions: Behavioral: Attention usual care
- Interactive advance care planning (Experimental): The intervention aims at facilitating patients, families, and primary physicians to discuss the patient's wishes for EOL care by clarifying a terminally ill cancer patient's understanding of his/her prognosis and treatment options and her/his readiness for engagement in ACP, appropriately weighting the benefits and burdens of medical treatments at EOL, and clearly defining and documenting the patient's preferences so as to be readily available later for the patient's primary physician to guide EOL care decision-making which will honor the patient's preferences for EOL care.
  Interventions: Behavioral: Interactive advance care planning

INTERVENTIONS:
Behavioral: Interactive advance care planning — The facilitator will begin each course of intervention by assessing the patient's and his/her family caregiver's readiness for engagement in ACP independently.
  Providing participant-centered care tailored to the specific needs of participants at each stage of readiness for engagement in ACP.
  Facilitating EOL care discussions throughout the dying process.
  A workbook and a video decision aid that briefly describes ACP to enhance participants' understanding of the essential elements in ACP.
  Other Names: Interactive ACP
  Arms: Interactive advance care planning
Behavioral: Attention usual care — a consistent master prepared nurse on the study team will provide the attention portion of the care. The initial meeting will occur before the patient discharges from hospital and the usual care nurse will give patients and family caregivers a workbook and a video with educational materials on how to manage common symptoms and a comprehensive list of resources available, including patient support organizations, support and financial assistance through the social work department..
  Arms: Attention usual care intervention

SUMMARY:
The purpose of this 5-year interventional study is to design, implement, and evaluate the effectiveness of an intervention aimed at facilitating prognosis communication and end-of-life care decision-making to increase the extent of congruence between the patient's preferred and actual EOL care received and patients' and family caregivers' QOL and psychological well-being, reduce futile aggressive healthcare resources utilization at end-of-life, and facilitate bereavement adjustment.

DETAILED DESCRIPTION:
A randomized controlled trial with a tailored, multifaceted intervention will be conducted on a convenience sample of 231 dyads of terminally ill cancer patients and caregivers with the same number of attention controlled group to evaluate the intervention's effectiveness.

Sample size calculation: There was no interventional study directly investigating the effectiveness in increasing the extent of congruence between patient preferred and actual end-of-life (EOL) care received by terminally ill cancer patients; therefore sample size estimation will be based on the effectiveness of holding EOL care discussions between patients and physicians on the extent to increase congruence between the patient's preferred and actual EOL care received. Patients who reported having EOL care discussions with their physicians significantly more likely to receive EOL care consistent to their preferences (OR=2.26; p<.0001) and received significantly fewer aggressive medical interventions near death, with lower rates of CPR (0.8% vs 6.7%; AOR, 0.16; 95% CI, 0.03-0.80), mechanical ventilation support (1.6% vs 11.0%; AOR, 0.26; 95% CI, 0.08-0.83), and ICU care (4.1% vs 12.4%; AOR, 0.35; 95% CI, 0.14-0.90), respectively. A sample size of 124-195 dyads per group achieves 80% power to detect a difference between the interventional and control group by a two-sided hypothesis test with a significance level of 0.05. In compensating the 18.5% of attrition rate found in our previous longitudinal study, 147-231 dyads per group are needed. The proposed sample size will be targeted on 231 dyads per group to ensure adequate power to detect the hypothesized effects of the proposed intervention.

Approximately 8-10 new dyads of terminally ill cancer patients and their family caregivers were recruited in each month. In order to recruit the targeted 462 dyads (231 dyads in each treatment group) of subjects, after development of detailed study protocol, subjects will start to enter into the study at the beginning of the 6th month of the study through the 54 th month and be followed through the 5th year of the proposed study period. We will enroll and randomly assign eligible dyads of terminally ill cancer patients and their family caregivers into intervention or attention controlled group in a 1:1 fashion without stratification.

Data collection procedures: Assessments will be performed prospectively and continue until patient death, loss to follow-up, study withdrawal, or when the patient can no longer be interviewed. An every-3-week time frame will be used in this study for repeated QOL and other outcomes assessments for both patients and their family caregivers bases on the review of literature to cover the most rapid change of patient physical conditions and demanding period of caregiving until the death of the patient. After each patient's death, a chart review and postmortem interview with patients' caregivers will be performed to confirm the type of medical care received at the EOL. Bereavement interviews will be conducted 1, 3, 6 and 13 months after the time of death in order to avoid contamination on the basis of anniversary grief reactions.1

Several strategies will be taken to ensure research fidelity.

1. The proposed intervention requires professionals skilled in the content, techniques, and delivery of the intervention. Built on her previous oncology and hospice care experiences, a competency-based educational approach will be used to train the facilitator. The training will include an overview of the study protocol and procedures, a review of the developed workbook and video, and instructions in motivational assessments. The principal investigator (PI) will serve as a role model for the facilitator to coach her how to assess and motivate participants at different stage of the readiness for engagement in ACP and cooperate with physicians in coordinating and facilitating EOL care discussions. The facilitator needs to successfully demonstrate predefined competencies and consistency to delivery of the ACP intervention after training and receipt of individual feedback from the PI before formal interventions can be conducted. Thereafter the study team will meet biweekly to review the facilitator's notes on interventional sessions and to provide feedback on difficult subject management issues.
2. Interventions provided to subjects assigned to the intervention group will be compared with those received by those who assigned to the control group every 3 months. Randomly selected dyads of terminally ill cancer patients and their family caregivers in each treatment group will be interviewed by the PI to check the extent to which treatments provided to them consistent with the protocol for each group.
3. To avoid bias, separate data collectors will be hired and trained for the study to collect data for the intervention and the control group independently. Training will include screening subjects, obtaining consents, and administering the project instruments without offering information; research assistants (RAs) will be blinded to treatment conditions. Procedures will be implemented to insure the standardization of data collection. RAs reliability will be established by comparing data collected by the RAs with that recorded by the PI on five pilot cases. Ninety-five percent agreements will be required before data collection for main study can begin. Failure to reach this agreement rate will require additional training until the acceptable reliability level is reached. Intermittent reliability checks will be carried out by the PI throughout the study to maintain a 95% agreement.
4. An independent Data and Safety Monitoring Board (DSMB) will be organized to ensure continuing patient safety as well as the validity and scientific merits of the trial. The DSMB will constitute a biostatistician experienced in statistical methods for clinical trials, a nursing researcher experienced in conducting RCTs, and a physician-scientist experienced in cancer care.

The DSMB will monitor and address the following issues: (1) sufficient and appropriate enrollment of subjects, including compliance with the eligibility criteria for each dyad of terminally ill cancer patients and family caregivers enrolled in the trial, (2) appropriate implementation of randomization, (3) comparability of baseline data between treatment groups, (4) protocol compliance, including treatments delivered to each treatment group and the data collection schemes,(5) adverse events (AEs), quality assurance for data validation and registry procedures for Clinical Trial registration at ClinicalTrials.gov.

A databet that records number of recruitment each month and the baseline information will be maintained to ensure sufficient and appropriate enrollment of subjects.

A dataset that captures the values the personnel used to randomize participants will be maintained, thereby allowing the process of treatment allocation to be reproduced and verified later. The DSMB will monitor the appropriate implementation of randomization by reviewing this dataset.

Interventions delivered to subjects assigned to the intervention and the attention-controlled group will be compared every 6 months by interviewing randomly selected dyads of terminally ill cancer patients and their family caregivers in each treatment group to check treatments provided to them.

AEs will be recorded and submitted by the study team in written to the DSMB monthly, with immediate reporting of serious AEs to the DSMB and an oncologist with expertise in cancer care. Site reports AEs/SAEs to its IRB will be dictated by local requirements.

No data will be analyzed before the study ended. Access to interim results, including results according to study arm will be limited to the DSMB members and the statistician who prepared the reports only. The DSMB will review study data every 6 months and the DSMB' summary recommendations will be directed to the PI. A summary of the review of reported AEs/SAEs will be sent to the local IRB to ensure that the participating center will be informed of any pertinent safety issues.

The biostatistician will be responsible for ensuring quality of data submitted to the registry against the predefined range of each independent and dependent variable and assessing the accuracy and completeness of registry data by comparing the submitted data to the original data.

Data analysis and interpretation:

1. All data will be scored and entered into a computer spreadsheet by an administrative assistant blinded to the group allocation of the participant.
2. In order to test for baseline group equivalence, differences between study groups in baseline characteristics and identified outcomes will be assessed with the use of two-sided Fisher's exact tests and chi-square tests for categorical variables and independent-samples Student's t-tests for continuous variables.
3. Intention-to-treat regression analyses will be performed with generalized estimating equations (GEE) to examine the effectiveness of intervention. In the intention- to-treat regression analyses, all participants will be analysed in the treatment group to which they are initially allocated regardless of whether they complete or withdraw from the treatment until the patient dies.
4. The extend of congruence of the terminally ill cancer patients' preferred and actual EOL care received will be obtained by comparing the agreement between the preferences of EOL care elicited at the last assessment and actual EOL care received by the patient by the percentage of overall agreement and kappa coefficients to assess the extent of congruence to correct for the amount of agreement that can be expected to occur by chance alone.
5. Multivariate logistic regression by the GEE will be used to examine the impact of intervention on improving the extend of congruence between terminally ill cancer patients' preferred and actual EOL care received, and secondary outcomes, namely increasing prognosis awareness, EOL care discussion, and the extent of patient-family agreement on preferences of EOL care, decreasing use of futile aggressive EOL care, and facilitating hospice use and early hospice referral, with simultaneously adjusting for confounding factors. The moderation effects of prognosis awareness, EOL care discussion, and patient-family agreement on preferences of EOL care on extend of congruence between terminally ill cancer patients' preferred and actual EOL care received, decreasing use of futile aggressive EOL care, and facilitating hospice use and early hospice referral between interventional group and the attention controlled group also will be examined in the GEE model.

7. Multivariate multiple regression by the GEE will be used to test the effectiveness of intervention in improving patients' and family caregivers' QOL and psychological well-being (anxiety and depression), and family bereavement outcomes (including QOL, depression, and grief reactions), with simultaneously adjusting for confounding factors. The moderation effects of prognosis awareness, EOL care discussion, and patient-family agreement on preferences of EOL care on the differences in patients' and family caregivers' QOL and psychological well-being before the patient's death, and family bereavement outcomes between intervention group and the attention controlled group also will be examined in the GEE model. How limiting futile aggressive EOL care and the extent of congruence between terminally ill cancer patients' preferred and actual EOL care received will moderate the intervention's effectiveness on improving patients' and family caregivers' QOL and psychological well-being before the patient's death and family bereavement outcomes also will be examined in the GEE model.

ELIGIBILITY:
Inclusion Criteria:

Terminally ill cancer patients are they:

1. have a disease at a terminal stage which continues to progress with distant metastases and is unresponsive to current curative cancer treatment as judged by their oncologists
2. are cognitively competent
3. can communicate with data collectors
4. age ≧ 20
5. have a designated family caregiver who agrees to participate in the survey.

Family caregivers will be recruited if they are:

1. family members of cancer patients with a terminally ill disease as defined by this proposed study
2. identified by the patients as the persons primarily conduct the patient's care needs without receiving financial reimbursement for the care they provide
3. age≧20
4. who agree to participate and can communicate with data collectors.

Exclusion Criteria:

1. Patients or family caregivers who are not able to communicate coherently.
2. Only one party in the patient-family dyad agrees to participate.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Congruence between preferred and actual EOL care received | An every-3-week time frame, at a minimum, after study enrollment until patient death or subject declining to participate will be used in this study for repeated outcomes assessments. Subjects will participate for an expected average of 5 months.
  EOL care includes (1) life-prolonging or comfort-oriented EOL care, (2) CPR when life is in danger, (3) life-sustaining treatments, including cardiac massage, mechanical ventilation, ICU care, tube feeding, intravenous nutrition, and hemodialysis, and (4) hospice care.
Quality of life for terminally ill cancer patients | An every-3-week time frame, at a minimum, after study enrollment until patient death or subject declining to participate will be used in this study for repeated outcomes assessments. Subjects will participate for an expected average of 5 months.
  McGill Quality of Life Questionnaire will be used to measure quality of life.
Psychological well-beings for terminally ill cancer patients | An every-3-week time frame, at a minimum, after study enrollment until patient death or subject declining to participate will be used in this study for repeated outcomes assessments. Subjects will participate for an expected average of 5 months.
  Depression and anxiety for terminally ill cancer patients.
  Anxiety and depressive symptoms of terminally ill cancer patients will be measured by the Hospital Anxiety and Depression Scale.
Family depressive symptoms | An every-3-week time frame, at a minimum, after study enrollment until patient death or subject declining to participate will be used in this study for repeated outcomes assessments. Subjects will participate for an expected average of 5 months.
  Depressive symptoms will be measured by the Center for Epidemiological Studies-Depression Scale.
Family quality of life | An every-3-week time frame, at a minimum, after study enrollment until patient death or subject declining to participate will be used in this study for repeated outcomes assessments. Subjects will participate for an expected average of 5 months.
  Quality of life for family caregivers while they provide end-of-life care will be measured by the Caregiver Quality of Life Index-Cancer.
Bereavement adjustment-Family depressive symptoms | Bereavement interviews will be conducted 1, 3, 6 and 13 months after the time of death in order to avoid contamination on the basis of anniversary grief reactions.
  Center for Epidemiological Studies-Depression Scale will be used to measure depressive symptom for bereaved family caregivers.
Bereavement adjustment-complicated grief | Bereavement interviews will be conducted 1, 3, 6 and 13 months after the time of death in order to avoid contamination on the basis of anniversary grief reactions.
  Complicated grief experience by family caregivers during their bereavement will be measured by the Inventory of Complicated Grief.

SECONDARY OUTCOMES:
Patient prognosis awareness | An every-3-week time frame, at a minimum, after study enrollment until patient death or subject declining to participate will be used in this study for repeated outcomes assessments. Subjects will participate for an expected average of 5 months.
  Terminally ill cancer patients' understanding whether their disease will be cured or not be cured and probability to die in the near future.
Family prognosis awareness | An every-3-week time frame, at a minimum, after study enrollment until patient death or subject declining to participate will be used in this study for repeated outcomes assessments. Subjects will participate for an expected average of 5 months.
  Family caregivers' understanding whether their relative's disease can be cured or not be cured and probability will die in the near future.
EOL care discussions among patients, families, and physicians | An every-3-week time frame, at a minimum, after study enrollment until patient death or subject declining to participate will be used in this study for repeated outcomes assessments. Subjects will participate for an expected average of 5 months.
  Discussions about the preferences for end-of-life care and advanced care planning.
The extent of patient-family agreement on the preferences of EOL care | An every-3-week time frame, at a minimum, after study enrollment until patient death or subject declining to participate will be used in this study for repeated outcomes assessments. Subjects will participate for an expected average of 5 months.
  The extent of patient-family agreements on preferences of cardiopulmonary resuscitation when life is in danger, life-sustaining treatments, including cardiac massage, mechanical ventilation, ICU care, tube feeding, intravenous nutrition, and hemodialysis, and hospice care.
Aggressive EOL care treatments | After each patient's death, a chart review and postmortem interview with patients' caregivers will be performed to confirm the type of medical care received at the EOL.
  Aggressive EOL care received by terminally ill cancer patients include cardiopulmonary resuscitation, life-sustaining treatments, including cardiac massage, mechanical ventilation, ICU care, tube feeding, intravenous nutrition, and hemodialysis, and hospice care.

CONTACTS AND LOCATIONS:
Overall Officials: Siew Tzuh Tang, DNSc, Principal Investigator — School of Nursing, Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital-LinKo, Linkou District, Taiwan

REFERENCES:
- [Background] Tang ST, Liu TW, Lai MS, Liu LN, Chen CH. Concordance of preferences for end-of-life care between terminally ill cancer patients and their family caregivers in Taiwan. J Pain Symptom Manage. 2005 Dec;30(6):510-8. doi: 10.1016/j.jpainsymman.2005.05.019. PMID 16376737
- [Background] Tang ST, Liu TW, Lai MS, McCorkle R. Discrepancy in the preferences of place of death between terminally ill cancer patients and their primary family caregivers in Taiwan. Soc Sci Med. 2005 Oct;61(7):1560-6. doi: 10.1016/j.socscimed.2005.02.006. Epub 2005 Apr 7. PMID 16005787
- [Background] Tang ST, Liu TW, Tsai CM, Wang CH, Chang GC, Liu LN. Patient awareness of prognosis, patient-family caregiver congruence on the preferred place of death, and caregiving burden of families contribute to the quality of life for terminally ill cancer patients in Taiwan. Psychooncology. 2008 Dec;17(12):1202-9. doi: 10.1002/pon.1343. PMID 18521969
- [Background] Tang ST, Wu SC, Hung YN, Huang EW, Chen JS, Liu TW. Trends in quality of end-of-life care for Taiwanese cancer patients who died in 2000-2006. Ann Oncol. 2009 Feb;20(2):343-8. doi: 10.1093/annonc/mdn602. Epub 2008 Sep 2. PMID 18765460
- [Background] Tang ST, Wu SC, Hung YN, Chen JS, Huang EW, Liu TW. Determinants of aggressive end-of-life care for Taiwanese cancer decedents, 2001 to 2006. J Clin Oncol. 2009 Sep 20;27(27):4613-8. doi: 10.1200/JCO.2008.20.5096. Epub 2009 Aug 24. PMID 19704067
- [Derived] Chen CH, Wen FH, Chang WC, Hsieh CH, Chou WC, Chen JS, Tang ST. Associations of prognostic-awareness-transition patterns with emotional distress and quality of life during terminally ill cancer patients' last 6 months of life. Psychooncology. 2023 May;32(5):741-750. doi: 10.1002/pon.6119. Epub 2023 Mar 14. PMID 36891618
- [Derived] Chen CH, Wen FH, Chou WC, Chen JS, Chang WC, Hsieh CH, Tang ST. Associations of prognostic-awareness-transition patterns with end-of-life care in cancer patients' last month. Support Care Cancer. 2022 Jul;30(7):5975-5989. doi: 10.1007/s00520-022-07007-4. Epub 2022 Apr 8. PMID 35391576
- [Derived] Wen FH, Chen CH, Chou WC, Chen JS, Chang WC, Hsieh CH, Tang ST. Evaluating if an Advance Care Planning Intervention Promotes Do-Not-Resuscitate Orders by Facilitating Accurate Prognostic Awareness. J Natl Compr Canc Netw. 2020 Dec 2;18(12):1658-1666. doi: 10.6004/jnccn.2020.7601. Print 2020 Dec. PMID 33285517
- [Derived] Wen FH, Chen JS, Chou WC, Chang WC, Hsieh CH, Tang ST. Extent and Determinants of Terminally Ill Cancer Patients' Concordance Between Preferred and Received Life-Sustaining Treatment States: An Advance Care Planning Randomized Trial in Taiwan. J Pain Symptom Manage. 2019 Jul;58(1):1-10.e10. doi: 10.1016/j.jpainsymman.2019.04.010. Epub 2019 Apr 18. PMID 31004770
- [Derived] Chen CH, Chen JS, Wen FH, Chang WC, Chou WC, Hsieh CH, Hou MM, Tang ST. An Individualized, Interactive Intervention Promotes Terminally Ill Cancer Patients' Prognostic Awareness and Reduces Cardiopulmonary Resuscitation Received in the Last Month of Life: Secondary Analysis of a Randomized Clinical Trial. J Pain Symptom Manage. 2019 Apr;57(4):705-714.e7. doi: 10.1016/j.jpainsymman.2019.01.002. Epub 2019 Jan 10. PMID 30639758

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT01912846/Prot_SAP_000.pdf